CLINICAL TRIAL: NCT07241091
Title: A Randomized Controlled Trial of High-Purity Type-I Collagen-Based Biomaterial (Surgicoll-Mesh®) as a Peritoneal Substitute to Prevent Post-Peritonectomy Complications in Patients Undergoing Cytoreductive Surgery
Brief Title: SurgiPerito Trial: High-Purity Type-I Collagen for Peritoneal Reconstruction After Cytoreductive Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adichunchanagiri Institute of Medical Sciences, B G Nagara (Other)
Collaborators: JSS Medical College Hospital (Unknown)
Responsible Party: Principal Investigator, Dr Naveen Narayan MS, MCh (Plastic Surgery), Professor & HoD, Department of Plastic Reconstructive & Aesthetic Surgery, Adichunchanagiri Institute of Medical Sciences, B G Nagara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIMS/IEC/266/2025
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Peritoneal Surface Malignancy; Postoperative Adhesion; Bowel Obstruction; Wound Complications; Surgical Site Infection After Major Surgery; Ovarian Cancer (OvCa)
Keywords: High-Purity Type-I Collagen; Collagen Biomaterial; Peritonectomy; Cytoreductive Surgery (CRS); Peritoneal Substitute; Adhesion Prevention; Peritoneal Reconstruction; Regenerative Collagen Matrix; HIPEC (Hyperthermic Intraperitoneal Chemotherapy); Intra-abdominal Healing
MeSH Terms: conditions — Peritoneal Neoplasms; Intestinal Obstruction; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Purity Type-I Collagen-based Peritoneal Substitute (Active Comparator): Patients undergoing cytoreductive surgery (CRS) with peritonectomy will receive intraoperative peritoneal reconstruction using High Purity Type-I Collagen-based Peritoneal Substitute, a sterile, resorbable, high-purity Type-I collagen biomaterial. The mesh is tailored to the peritonectomy defect and secured with absorbable sutures prior to abdominal closure.
  Interventions: Device: High-Purity Type-I Collagen Scaffold
- Standard Peritonectomy Closure (Active Comparator): Patients undergoing cytoreductive surgery with peritonectomy will have standard closure of the peritoneal defect without the use of any biomaterial or mesh substitute. Surgical closure will follow institutional standard of care.
  Interventions: Procedure: Standard Peritonectomy Closure

INTERVENTIONS:
Device: High-Purity Type-I Collagen Scaffold — Peritoneal reconstruction using High-Purity Type-I Collagen Scaffold after peritonectomy. Purpose is to act as a biologic peritoneal substitute promoting tissue regeneration and reducing postoperative adhesions and complications.
  Arms: High Purity Type-I Collagen-based Peritoneal Substitute
Procedure: Standard Peritonectomy Closure — Conventional Closure, to serve as the comparator arm for evaluating complication rates, adhesion formation, and recovery outcomes.
  Arms: Standard Peritonectomy Closure

SUMMARY:
This dual-centre, randomized controlled trial evaluates the safety and efficacy of high-purity Type-I collagen-based biomaterial, as a peritoneal substitute following peritonectomy in patients undergoing cytoreductive surgery (CRS) for peritoneal surface malignancy. The study tests whether Surgicoll-Mesh can reduce major postoperative intra-abdominal complications compared with standard management.

DETAILED DESCRIPTION:
Peritonectomy during CRS often leads to adhesion formation, obstruction, and wound complications. High-purity Type-I collagen-based biomaterial, a resorbable collagen matrix, provides a temporary barrier and scaffold that promotes tissue regeneration and reduces adhesions. This trial will randomize 60 patients (30 per group) to receive standard closure or peritoneal reconstruction with high-purity Type-I collagen-based biomaterial. The primary endpoint is the incidence of major intra-abdominal complications within 2 months. Secondary endpoints include individual complication rates, bowel recovery, hospital stay, mesh-related events, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosed peritoneal surface malignancy (colorectal, ovarian, appendiceal, mesothelioma, pseudomyxoma)
* Undergoing cytoreductive surgery ± HIPEC requiring peritonectomy
* ECOG 0-2, adequate organ function, informed consent

Exclusion Criteria:

* Collagen allergy or active infection
* Immunosuppression or chronic steroid use
* Pregnancy/lactation
* Uncontrolled sepsis, bowel perforation, or extensive small bowel resection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of major intra-abdominal complications | 2 months post-surgery
  Incidence of major intra-abdominal complications (adhesive SBO, enterocutaneous fistula, reoperation, grade ≥3 wound complication) within 2 months post-surgery

SECONDARY OUTCOMES:
Individual complication rates | 2 months
  Individual complication rates (intraperitoneal adhesions, bowel obstruction, wound infection, hernia, fistula)
Time to bowel function recovery | 1 month
  Time to bowel function recovery and diet tolerance
Length of hospital and ICU stay | 2 months
  Duration (in days) from the date of surgery until discharge from the hospital, including the number of days spent in the ICU. This will capture differences in postoperative recovery and resource utilization between groups.
Device-related adverse events | 2 months
  Any adverse event deemed related to the implanted High-Purity Type-I Collagen biomaterial, including mesh reaction, infection, seroma, rejection, or need for mesh removal, assessed within the 2-month postoperative period.
Quality of life Assessment | 2 months
  Quality of life assessment using the European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The questionnaire includes multiple subscales scored from 0 to 100. For functional scales and global health status, higher scores indicate better quality of life; for symptom scales, higher scores indicate worse symptoms.
Number of participants with MRI-detected intra-abdominal adhesions or obstruction | 2 months
  Radiologic assessment of intra-abdominal adhesions, bowel obstruction, or other postoperative abnormalities on MRI at baseline, 1 month, and 2 months. The number of participants demonstrating each finding will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: NAVEEN NARAYAN, MS, MCh, Study Chair — Adichunchanagiri Institute of Medical Sciences
Locations (2):
- India (2):
  - Adichunchanagiri Institute of Medical Sciences, Mandya, Karnataka
  - JSS Medical College Hospital, Mysore, Karnataka

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and statistical code will be available upon reasonable request after publication of results.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months post-publication
Access Criteria: De-identified individual participant data will be made available to investigators upon reasonable request beginning 6 months after publication. Access will be granted to researchers who provide a methodologically sound proposal and agree to use the data only for research purposes. Researchers must sign a data access agreement. The Study Protocol and Statistical Analysis Plan (SAP) will also be shared 6 months post-publication.

REFERENCES:
- [Background] Naveen Narayan, KN rajeSh, ChethaN ShivaNNaiah, SuhaS N Gowda. Collagen-based Mesh in the Treatment of Posthernioplasty Mesh Infection in Ventral Hernias: A Case Series. Journal of Clinical and Diagnostic Research. 2024 Sep, Vol-18(9): PR01-PR03
- [Background] Narayan N, Gowda S, Shivannaiah C. A Randomized Controlled Clinical Trial Comparing the Use of High Purity Type-I Collagen-Based Skin Substitute vs. Dehydrated Human Amnion/Chorion Membrane in the Treatment of Diabetic Foot Ulcers. Cureus. 2024 Dec 5;16(12):e75182. doi: 10.7759/cureus.75182. eCollection 2024 Dec. PMID 39649230
- [Background] Narayan N, Shivannaiah C, Gowda S. Evaluating the Efficacy of High-Purity Type I Collagen-Based Skin Substitute Versus Dehydrated Human Amnion/Chorion Membrane in the Treatment of Venous Leg Ulcers: A Randomized Controlled Clinical Trial. Cureus. 2025 Jul 30;17(7):e89031. doi: 10.7759/cureus.89031. eCollection 2025 Jul. PMID 40747200
- [Background] Narayan N, Ramegowda YH, Raghupathi DS, Chethan S, Gowda S. Biological Skin Substitutes in Pressure Ulcers: High-Purity Type I Collagen-Based Versus Amnion/Chorion Membrane. Cureus. 2025 Aug 25;17(8):e90956. doi: 10.7759/cureus.90956. eCollection 2025 Aug. PMID 40862036
- [Background] Dhanraj P, Naveen N, Babu KR, Mahesh M, Hanumanthaiah KS: Healicoll - an alternate to flap cover for bare bones and tendons. Acta Medica International. 2016, 3:146-50.
- [Background] Naveen N, Dharini K, Yashas HR: Multifaceted role of the acellular dermal matrix in novel wound healing: a case series. J Clin Diag Res. 2025, 19:01-05. 10.7860/JCDR/2025/79891.21070
- [Background] Subramanian A, Liang MK. A 60-year literature review of stump appendicitis: the need for a critical view. Am J Surg. 2012 Apr;203(4):503-7. doi: 10.1016/j.amjsurg.2011.04.009. Epub 2011 Dec 6. PMID 22153086
- [Background] Tzivanakis A, Dayal SP, Arnold SJ, Mohamed F, Cecil TD, Venkatasubramaniam AK, Moran BJ. Biological mesh is a safe and effective method of abdominal wall reconstruction in cytoreductive surgery for peritoneal malignancy. BJS Open. 2018 Aug 2;2(6):464-469. doi: 10.1002/bjs5.93. eCollection 2018 Dec. PMID 30511047